CLINICAL TRIAL: NCT05363215
Title: A Phase 1, Open-label, Parallel-group Study to Assess the Pharmacokinetics, Safety, and Tolerability of S-217622 in Participants With Mild, Moderate, and Severe Renal Impairment and Healthy Control Participants
Brief Title: A Study to Assess S-217622 in Participants With Renal Impairment and Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2128T1214
Record Dates: First submitted 2022-05-03; First posted 2022-05-05 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — ensitrelvir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- S-217622: Group A (Experimental): Participants with mild renal impairment will receive a single dose of S-217622 on Day 1, in a fasted state.
  Interventions: Drug: S-217622
- S-217622: Group B (Experimental): Participants with moderate renal impairment will receive a single dose of S-217622 on Day 1, in a fasted state.
  Interventions: Drug: S-217622
- S-217622: Group C (Experimental): Participants with severe renal impairment will receive a single dose of S-217622 on Day 1, in a fasted state.
  Interventions: Drug: S-217622
- S-217622: Group D (Experimental): Participants with normal renal function will receive a single dose of S-217622 on Day 1, in a fasted state.
  Interventions: Drug: S-217622

INTERVENTIONS:
Drug: S-217622 — Tablet for oral administration

SUMMARY:
The objective of this study is to measure the PK, safety, and tolerability of S-217622 in participants with mild, moderate, or severe renal impairment and in those with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 50 kilograms (kg) and body mass index (BMI) within the range of ≥ 18.5 to < 38.0 kilogram-meter squared (kg/m^2) at the Screening visit

Participants With Renal Impairment

* Participants that are not undergoing dialysis must have mild, moderate, or severe renal impairment based upon their Modification of Diet in Renal Disease (MDRD) creatinine clearance estimate (estimated glomerular filtration rate [eGFR]) calculated at the Screening visit:

  1. Mild renal impairment: 60 to 89 milliliters per minute (mL/min)/1.73 m^2
  2. Moderate renal impairment: 30 to 59 mL/min/1.73 m^2
  3. Severe renal impairment: No lower limit of eGFR, <30 mL/min
* A stable medication regimen is required, defined as not starting new drug(s) or changing dosage(s) within 14 days prior to administration of study intervention through the Follow-up/Early Termination visit.

Healthy Participants

* Participants with clinical laboratory tests within normal reference range for the laboratory, or abnormal but considered not clinically significant by the investigator. Renal function, calculated by MDRD, must be normal (ie, eGFR > 90 mL/min/1.73 m^2).
* Matched to each participant with moderate renal impairment with respect to sex, age (± 5 years), and BMI (± 10%).

Exclusion Criteria:

* Participants with life expectancy less than 3 months.
* History or presence of/significant history of or current cardiovascular, respiratory, hepatic, gastrointestinal (GI), endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of GI surgery including but not limited to gastric resection and/or intestinal resection that resulted in a clinically significant abnormality in GI function.
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Breast cancer within the past 10 years.
* Participant with poor venous access.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of S-217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15
Time to Maximum Plasma Concentration (Tmax) of S-217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15
Area Under the Plasma Concentration-Time Curve (AUC) of S-217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15
Terminal Elimination Half-Life (t1/2,z) of S-217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15
Terminal Elimination Rate Constant (λz) of S-217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15
Mean Residence Time (MRT) of S-217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15
Apparent Total Clearance (CL/F) of S-217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15
Apparent Volume of Distribution (Vz/F) of S-217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15
Renal Clearance (CLR) of S-217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15
Fraction of Dose Excreted in Urine (Feu) of S-217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15
Fraction Unbound in Plasma (FU) of S217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15

SECONDARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events | Up to Day 21

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Orlando Clinical Research Center, Inc., Orlando, Florida
  - Nucleus Network, Saint Paul, Minnesota